CLINICAL TRIAL: NCT06889454
Title: The Effect of Different Treatment Options on Markers of Vascular, Myocardial and Endothelial Function in Women With Polycystic Ovary Syndrome and the Association With Metabolic and Hormonal Abnormalities of the Syndrome
Brief Title: Cardiovascular and Endothelial Markers During OGTT Before and at Six and Twelve Months Post-treatment in Women With PCOS
Status: Recruiting | Type: Observational
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, VAIA LAMBADIARI, Professor of Internal Medicine-Endocrinology, Attikon Hospital
Other Study IDs: PCOS_OGTT
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: PCOS; Hyperinsulinism; Hyperandrogenism; Metabolic Syndrome
MeSH Terms: conditions — Hyperinsulinism; Hyperandrogenism; Metabolic Syndrome | interventions — Contraceptives, Oral; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- GLP-1 agonists: 30 women will receive lifestyle modification and GLP-1RA.
  Interventions: Drug: GLP-1 receptor agonist
- Oral contraceprives: 30 women will receive lifestyle modification and OCP.
  Interventions: Drug: Oral contraceptive
- Metformin: 30 women will receive lifestyle modification and metformin
  Interventions: Drug: Metformin
- Lifestyle Modification: 30 women will receive only lifestyle modification
  Interventions: Other: Lifestyle modification

INTERVENTIONS:
Drug: GLP-1 receptor agonist — 30 women will receive lifestyle modification and GLP-1 receptor agonists
  Groups: GLP-1 agonists
Drug: Oral contraceptive — 30 women will receive lifestyle modification and oral contraceptive
  Groups: Oral contraceprives
Drug: Metformin — 30 women will receive lifestyle modification and metformin
  Groups: Metformin
Other: Lifestyle modification — 30 women will receive only lifestyle modification
  Groups: Lifestyle Modification

SUMMARY:
The aim of the present study is to investigate a) the presence of subclinical markers of vascular, myocardial and endothelial function in women with PCOS b) the acute alterations in these markers during the oral glucose tolerance test (OGTT) c) the impact of potential treatment interventions in these markers.

DETAILED DESCRIPTION:
All the woman who will recruited in the study will undergo OGTT. At 0, 60, and 120 min of glucose load the investigators will measure: a) glucose and insulin, b) pulse wave velocity (PWV) c) augmentation index (Aix) and d) perfused boundary region of sublingual microvessels (high PBR values represent reduced glycocalyx thickness). At 0 and 120 min of glucose load, the investigators will assess: a) coronary flow reserve (CFR) using Doppler echocardiography, b) LV longitudinal strain (LS) of subendocardial, mid-myocardial and subepicardial layers and global LS (GLS) c) peak twisting (pTw), untwisting velocity (pUtwVel) by speckle tracking echocardiography d) flow mediated dilation (FMD) of the brachial artery, e) Carotid intima-media thickness. Matsuda index, insulin sensitivity index (ISI) and HOMA index will be also measured. The levels of Testosterone (Τesto), Sex hormone binding globulin (SHBG), dehydroepiandrosterone sulfate (DHEA-s), Prolactin (PRL), 17-hydroxyprogesterone (17-OH-PRG) ,Androstenedione (Δ4) and Metalloproteinase 9 will be also assessed. After six months of treatment intervention, the patient will undergo the previously described measurements. Primary Endpoints include the change in GLS, PWV, and PBR during OGTT and six months after treatment intervention. Secondary Endpoints include the change in CFR and FMD during OGTT and six months after treatment intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 16 years old
2. Diagonis of PCOS according to Rotterdam criteria: presence of two of the three of the following:

   * Clinical or biochemical hyperandrogenism
   * Anovulation or oligo-ovulation
   * Polycystic ovarian morphology (PCOM)
3. Absence of treatment for PCOS the last six months
4. Patients who have the ability to understand and sign the consent form.

Exclusion Criteria:

1. Disorders with clinical presentation similar to PCOS: thyroid disease, hyperprolactinemia, and non-classic congenital adrenal hyperplasia (primarily 21-hydroxylase deficiency by serum 17-hydroxyprogesterone [17-OHP]), Cushing syndrome, acromegaly
2. Treatment with contraceptive or metformin
3. Type 2 diabetes mellitus
4. Treatment for diabetes
5. Pregnancy
6. Lactation
7. Malignancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with PCOS
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Τhe change in Global Longitudinal Strain during Oral glucose Tolerance Test | 120 minute of Oral glucose Tolerance Test
  Τhe change in Global Longitudinal Strain at 0 and 120 minute after glucose load
The change in Pulse Wave Velocity during Oral glucose Tolerance Test | 120minute of Oral glucose Tolerance Test
  The change in Pulse Wave Velocity at 0 and 120 minute after glucose load
The change in Perfused Boundary Region during Oral glucose Tolerance Test | 120minute of Oral glucose Tolerance Test
  The change in Perfused Boundary Region at 0 and 120 minute after glucose load
The change in Global Longitudinal Strain | six months
  The change in Global Longitudinal Strain 6 months after treatment intervention
The change in Pulse Wave Velocity | six months
  The change in Pulse Wave Velocity 6 months after treatment intervention
The change in Perfused Boundary Region | six months
  The change in Perfused Boundary Region 6 months after treatment intervention
The change in Metalloproteinase 9 | six months
  The change in Metalloproteinase 9 six months after tretament intervention

SECONDARY OUTCOMES:
Τhe change in Coronary flow reserve during Oral glucose Tolerance Test | 120 min of Oral glucose Tolerance Test
  Τhe change in Coronary flow reserve at 0 and 120 min after glucose load
Τhe change in Flow mediated Dilation during Oral glucose Tolerance Test | 120min of Oral glucose Tolerance Test
  Τhe change in Flow mediated Dilation at 0 and 120 min after glucose load
The change in Coronary flow reserve | six months
  The change in Coronary flow reserve 6 months after treatment intervention
The change in Flow mediated Dilation | six months
  The change in Flow mediated Dilation 6 months after treatment intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon University General Hospital, Chaïdári, Greece

IPD SHARING:
Plan to Share IPD: Undecided